CLINICAL TRIAL: NCT05386758
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Molnupiravir (MK-4482; MOV) in Participants With Severe Renal Impairment
Brief Title: A Study to Evaluate Molnupiravir (MK-4482; MOV) in Participants With Severe Renal Impairment (MK-4482-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4482-003; MK-4482-003 (Other: MSD)
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — molnupiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel A - Severe Renal Impairment Group (Experimental): Participants with severe renal impairment will receive a single oral 800 mg dose of molnupiravir.
  Interventions: Drug: Molnupiravir
- Panel B - Healthy Control Group (Experimental): Participants in the healthy mean matched control group will receive a single oral 800 mg dose of molnupiravir.
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Molnupiravir — Four 200 mg capsules administered orally as a single dose
  Other Names: MK-4482; MOV; EIDD-2801

SUMMARY:
This purpose of this study is to evaluate the plasma pharmacokinetics (PK) of N-hydroxycytidine (NHC), the nucleoside metabolite of molnupiravir, after a single oral dose of 800 mg molnupiravir in participants with severe renal impairment compared to healthy mean matched control participants. This study will also assess the safety and tolerability of molnupiravir in participants with severe renal impairment and the urinary excretion of NHC after a single oral dose of 800 mg molnupiravir in participants with severe renal impairment compared to healthy mean matched control participants. The primary hypothesis is that the plasma PK participants with severe renal impairment will be similar to that observed in the healthy mean matched control participants.

ELIGIBILITY:
Inclusion Criteria:

The key Inclusion Criteria include but are not limited to the following:

* Body mass index (BMI) ≥18.5 kg/m^2 and ≤35 kg/m^2
* Healthy participants: Baseline estimated glomerular filtration rate (eGFR) ≥90 mL/min based on the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine equation
* Severe renal impairment participants: Baseline estimated glomerular filtration rate (eGFR) <30 mL/min based on the 2021 CKD-EPI Creatinine equation

Exclusion Criteria:

The key Exclusion Criteria include but are not limited to the following:

* Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)
* History of major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit

Severe renal impairment participants:

* History or presence of renal artery stenosis
* Had a renal transplant
* Currently taking medications to treat chronic medical conditions associated with renal disease if participant has not been on a stable regimen for at least 1 month and/or is unable to withhold the use of medication(s) within 4 hours prior to and 8 hours after administration of the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Velocity Clinical Research, Hallandale Beach ( Site 0005), Hallandale, Florida
  - Advanced Pharma CR, LLC ( Site 0004), Miami, Florida
  - Genesis Clinical Research, LLC ( Site 0003), Tampa, Florida
  - Thomas Jefferson University-Pharmacology, Physiology and Cancer Biology ( Site 0001), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Duncan KE, Carstens RP, Butterfield KL, Jin Y, Inbody LR, Schaeffer AK, Matthews CZ, Zhao T, Patel S, Maas BM, Cheng MH, Stoch SA. Assessment of pharmacokinetics and tolerability following single-dose administration of molnupiravir in participants with hepatic or renal impairment. Clin Transl Sci. 2024 Dec;17(12):e70073. doi: 10.1111/cts.70073. PMID 39601078
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Severe Renal Impairment: Participants with severe renal impairment received a single oral 800 mg dose of molnupiravir.
- Healthy Participants With Normal Renal Function: Participants in the healthy mean matched control group received a single oral 800 mg dose of molnupiravir.
Period: Overall Study
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (7.9) | 59.6 (2.0) | 61.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of N-hydroxycytidine (NHC)
Description: Blood for plasma samples was collected at pre-specified time points to determine the AUC0-inf of NHC.
Time Frame: Predose, 0.5,1.5, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose
Population: All participants who complied with the protocol sufficiently to ensure that generated data likely exhibiting the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Number analyzed (Participants) | 8 | 8
hr*ng/mL | 11100 [7990 to 15400] | 8960 [7660 to 10500]
Statistical Analysis 1: Comparison: Participants With Severe Renal Impairment vs Healthy Participants With Normal Renal Function; Test type: Other; Gemetric Mean Ratio (GMR) = 1.24, 90% CI 2-sided [0.94 to 1.64]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of NHC
Description: Blood for plasma samples was collected at pre-specified time points to determine the Cmax of NHC.
Time Frame: Predose, 0.5,1.5, 2, 4, 6, 8, 12, 24, 48 and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Number analyzed (Participants) | 8 | 8
ng/mL | 3920 [2810 to 5460] | 3240 [2630 to 4000]
Statistical Analysis 1: Comparison: Participants With Severe Renal Impairment vs Healthy Participants With Normal Renal Function; Test type: Other; Geometric Mean Ratio (GMR) = 1.21, 90% CI 2-sided [0.90 to 1.62]

3. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was therefore any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE were reported.
Time Frame: Up to Day 15
Population: All participants who received at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants | 2 | 0

4. Secondary Outcome: Amount of Dose Administered Excreted in Urine (Ae) of N-hydroxycytidine (NHC)
Description: Urine was collected at pre-specified time points to determine the amount of dose Administered excreted in urine (Ae) of NHC.
Time Frame: Predose, 4, 8, 12 and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Number analyzed (Participants) | 8 | 8
mg | 3.72 (50.9) | 14.6 (172)

5. Secondary Outcome: Fraction of the Dose Administered Excreted in Urine (Fe) of NHC
Description: Urine was collected at pre-specified time points to determine the Fraction of the dose administered excreted in urine (Fe) of NHC.
Time Frame: Predose, 4, 8, 12 and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of administered dose
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Number analyzed (Participants) | 8 | 8
% of administered dose | 0.591 (50.9) | 2.33 (172)

6. Secondary Outcome: Renal Clearance (CLr) of NHC
Description: Urine will be collected at pre-specified time points to determine the Renal Clearance (CLr) of NHC
Time Frame: Predose, 4, 8, 12 and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
Number analyzed (Participants) | 8 | 8
L/hr | 0.338 (62.1) | 1.64 (162)

ADVERSE EVENTS:
Time Frame: Up to ~ Day 15
Description: All-cause mortality (ACM) was analyzed in all allocated participants. Safety Analyses were conducted in all participants who received at least 1 dose of study intervention.
Arm/Group | Participants With Severe Renal Impairment | Healthy Participants With Normal Renal Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Renal Impairment (N=8) | Healthy Participants With Normal Renal Function (N=8)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT05386758/Prot_SAP_000.pdf